CLINICAL TRIAL: NCT05073965
Title: Vitamin D Supplementation Effect In Children With Pulmonary Tuberculosis Treatment: Randomized Double Blind Controlled Trial
Brief Title: Vitamin D Supplementation Effect In Children With Pulmonary Tuberculosis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Lianda Tamara, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Paed-202108.01
Record Dates: First submitted 2021-08-27; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Subject receive a 1000IU vitamin D supplement dose daily for 6 months
  Interventions: Dietary Supplement: Vitamin D
- Placebo group (Placebo Comparator): Subject receive a placebo daily for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Subjects were assigned to receive a 1000IU vitamin D supplement dose
  Arms: Intervention Group
Other: Placebo — Subject were assigned to receive a placebo
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the vitamin D supplementation effect to improve clinical outcomes in children with pulmonary tuberculosis treatment. This randomized, double-blind control trial with a cohort design was conducted in West Borneo from December 2020 - July 2021. A Total 84 patients met the inclusion criteria; aged 6 to 18 years old, newly diagnosed with pulmonary tuberculosis with vitamin D insufficiency. Only 80 patients completed the six months follow-up. The intervention was 1,000 IU vitamin D or placebo for six months treatment. Comparison of clinical conditions and nutritional status are analyzed statistically.

DETAILED DESCRIPTION:
This randomized, double-blind control trial with a cohort design was conducted in Bethesda Hospital West Borneo from December 2020 - May 2021. The inclusion criteria were children between 6 to 18 years old, newly diagnosed with pulmonary tuberculosis with vitamin D insufficiency. Diagnosis of the tuberculosis case was based on The Indonesian Pediatric Tuberculosis Scoring System. It consists of history taking and laboratory findings that support tuberculosis common symptoms such as household contact, prolonged fever more than two weeks, non-remitting cough more than three weeks, and decrease body weight, and lymph node enlargement; laboratory findings include Tuberculin Skin Test (TST) and chest X-ray (CXR). Scoring ranges from 0 to 3 for each variable with a total score of more than six is considered as tuberculosis diagnosis. Patients also collect the sputum for gram staining and Xpert MTB/RIF examination. The isolation of Mycobacterium tuberculosis was not done in this study because of limited resources.

Subject selection was determined based on consecutive sampling, namely the order of patients who came to the clinic until the minimum sample size (84 subjects) met the inclusion criteria. The investigators excluded children with a history of liver or kidney abnormalities, immunocompromised, and already received vitamin D supplementation. After obtaining written consent, all subjects had their blood specimens drawn 3cc from the brachial vein to measure alanine transaminase (ALT), alkaline phosphatase (ALP), serum active 25-hydroxyvitamin D using the ELISA method. Vitamin D is categorized as deficiency if serum 25-hydroxyvitamin D is below 20ng/mL, insufficiency between 20-30ng/mL, and normal levels above 30ng/mL. In this study, the 95% confidence level (Zα = 1.65 one-sided test) and 80% power test (Zß = 0.84) were selected. The calculation of the sample size above obtained n = 35 people for each group. The total study subjects were added by 20% of the minimum number of samples to compensate for loss-to-follow-up, so the total sample was 84, consisting of 42 patients in the intervention group and 42 patients in the placebo group.

For each subject, the following data were entered into the study database demographic data ( name, age, sex), signs and symptoms (fever, cough), Tuberculin Skin Test (TST), Chest X-Ray, and also GeneXpert for Mycobacterium tuberculosis from gastric lavage or sputum induction, liver function test and 25-hydroxyvitamin D level. All results were recorded in a study database following international standards to protect the privacy and personal information.

Subjects were randomly assigned to receive either a 1000IU vitamin D supplement dose or a placebo with an allocation ratio of one to one. Before starting recruitment, the project manager prepared 84 packs of study preparation - 42 packs of the active study drug and 42 packs of a placebo, then generated a randomization sequence using a computer program assigning the terms active or placebo to numbers 1 to 84. The packs were then assigned a randomized number according to this computer-generated randomization sequence.

At recruitment, study staff enrolled patients consecutively according to the order of arrival of patients from number 1 to 84. Study staff who assigned patients to active drugs or placebo did not know the following assignment in the sequence because they did not have access to the study code. Treatment allocations were hidden from patients and research staff. Those who analyzed the data were not covered for group assignments. Monitoring of subjects medication adherence and daily symptoms conducted by using a checklist table filled out by the patient's parents and confirmed check by the researcher during the patient follow-up schedule to the clinic.

All subjects received antimicrobial treatment for tuberculosis drugs in the form of a fixed-dose combination. Patients were reviewed monthly after starting antimicrobial treatment; body weight and height were measured at each time point. After the intensive phase of antimicrobial treatment, patients were monitored monthly. A repeated vitamin D level by ELISA and liver function test were done six months after starting the antimicrobial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 18 years old
* Newly diagnosed with pulmonary tuberculosis
* Vitamin D insufficiency

Exclusion Criteria:

* Children with a history of liver abnormalities
* Children with a history of kidney abnormalities
* Immunocompromised children
* Children who has already received vitamin D supplementation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Cough Symptom | Baseline, every month in month 1-6
  Resolution time for coughing, parents take notes every day.
Change in Fever Symptom | Baseline, every month in month 1-6
  Resolution time for fever, parents take notes every day.
Change in Body weight | Baseline, every 2 weeks in month 1 and month 2, every month in month 3-6.
  Measurement of body weight
Change in Height | Baseline, every 2 weeks in month 1 and month 2, every month in month 3-6.
  Measurement of height
Change in Body Mass Index | Baseline, every 2 weeks in month 1 and month 2, every month in month 3-6.
  Calculation of Body Mass Index

SECONDARY OUTCOMES:
Vitamin D level | Baseline and 6 months after intervention
  Measurement of 25-hydroxyvitamin D serum level
Alanine Transaminase | Baseline and 6 months after intervention
  Measurement of alanine transaminase (ALT) serum level
Alkaline Phosphatase | Baseline and 6 months after intervention
  Measurement of alkaline phosphatase (ALP) serum level

CONTACTS AND LOCATIONS:
Overall Officials: Lianda Tamara, MD,Paed, Principal Investigator — Universitas Padjadjaran
Locations (1):
- RS Bethesda, Bengkayang, West Borneo, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamara L, Kartasasmita CB, Alam A, Gurnida DA. Effects of Vitamin D supplementation on resolution of fever and cough in children with pulmonary tuberculosis: A randomized double-blind controlled trial in Indonesia. J Glob Health. 2022 Feb 18;12:04015. doi: 10.7189/jogh.12.04015. eCollection 2022. PMID 35198149

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT05073965/Prot_ICF_000.pdf